CLINICAL TRIAL: NCT01089452
Title: ACCESS STUDY (Angiotensin Receptor Blocker Combined With Calcium Antagonist Evaluation of Safety and Lowering of Systolic Blood Pressure Study) ARB/CCB Combination Therapy: Efficacy vs an ACE-inhibitor/CCB Combination and Use as First Line Therapy.
Brief Title: Angiotensin Receptor Blocker Combined With Calcium Antagonist Evaluation of Safety and Lowering of Systolic Blood Pressure Study
Acronym: ACCESS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study not started due to administrative reasons.
Sponsor: Monash University (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Prof Henry Krum, Monash University / Alfred Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-01/09; HREC/10/Alfred/5 (Other: Consultative Council for Human Research Ethics); 62/10 (Other: Alfred Hospital)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
Keywords: Mild to moderate hypertension
MeSH Terms: conditions — Hypertension | interventions — Perindopril; amlodipine, perindopril drug combination; olmesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perindopril monotherapy (Active Comparator): Perindopril 5mg for 4 weeks, forced titration to 10mg for 8 weeks
  Interventions: Drug: Perindopril
- Perindopril/amlodipine (Active Comparator): Perindopril/amlodipine 5/5mg, 10/5mg, 10/10mg: 4 weeks duration at each dose; forced titration.
  Interventions: Drug: Perindopril/amlodipine
- Olmesartan/amlodipine FDC (Experimental): Olmesartan/amlodipine 20/5mg, 40/5mg, 40/10mg: 4 weeks at each dose; forced titration.
  Interventions: Drug: Olmesartan/amlodipine

INTERVENTIONS:
Drug: Perindopril — Perindopril 5mg for 4 weeks, forced titration to 10mg for 8 weeks
  Arms: Perindopril monotherapy
Drug: Perindopril/amlodipine — Perindopril/amlodipine 5/5mg, 10/5mg, 10/10mg: 4 weeks duration at each dose; forced titration.
  Arms: Perindopril/amlodipine
Drug: Olmesartan/amlodipine — Olmesartan/amlodipine 20/5mg, 40/5mg, 40/10mg: 4 weeks at each dose; forced titration.
  Arms: Olmesartan/amlodipine FDC

SUMMARY:
This study is looking to evaluate which drug combination, olmesartan/amlodipine or perindopril/amlodipine, is better at lowering blood pressure in people with mild to moderate hypertension. The investigators will be enrolling people who are either currently taking medication to lower their blood pressure or who have been recently diagnosed with high blood pressure and are not yet on medication.

Patients on medication for their blood pressure will be asked to stop taking this medication for 2 to 4 weeks. If their blood pressure is suitable (not too high or low) they will be randomised to one of their treatment arm:

Group 1 will receive Perindopril on its own (5mg for 4 weeks followed by 10mg for 8 weeks). There will be 80 patients in this group.

Group 2 will receive Perindopril and Amlodipine together (5mg/5mg for 4 weeks, 10mg/5mg for a further 4 weeks then 10mg/10mg for the final 4 weeks). There will be 80 patient in this group.

Group 3 will receive Olmesartan and Amlodipine together (20mg/5mg for 4 weeks, 40mg/5mg for a further 4 weeks then 40mg/10mg for the final 4 weeks). There will be 120 patients in this group.

During the study we will measure the patients blood pressure and heart rate, weight and perform routine blood tests. They will also have ECGs (3 occasions) and 24 hour blood pressure monitor (4 occasions).

At the end of the study patients pre-study medication will be restarted or they will be put on to a suitable alternative.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Has provided written informed consent
3. Mild to moderate hypertension (WHO Stage 1-2). Patients with mild to moderate hypertension will be either de novo presenters with this condition or withdrawn from background antihypertensive therapy for a period of 2 weeks. If sSBP is not greater than 140 mmHg after this 2 week withdrawal period (*130 mmHg if diabetes or CKD, as per Heart Foundation of Australia Hypertension Guidelines 20082), patients can be followed, off therapy, for a further 2 weeks in order to meet this criterion. If their systolic blood pressure is above 180 mmHg they will be withdrawn from the study and will be provided with appropriate treatment.
4. Hypertensive patients with a high level of risk, i.e. having at least one of the following risk factors :

   * History of CV event eg MI, stroke (>6 months ago)
   * History of revascularization procedure (>6 months ago)
   * Impaired kidney function (eGFR <70 ml/min)
   * ECG or echocardiographic evidence of LV hypertrophy
   * Obesity, defined as BMI >30 kg/m2
   * Diabetes mellitus
   * Peripheral arterial disease
   * Macroalbuminuria
   * Current smoking (defined as smoking at least 7 cigarettes per week)
5. Women must be post menopausal or using an acceptable method of contraception i.e. surgical sterilisation, hormonal contraception or double barrier method.

Exclusion Criteria:

1. Secondary causes of hypertension (e.g. Conn's Syndrome, renal artery stenosis)
2. Serum creatinine >0.25 mmol/L or eGFR <40 ml/min
3. Serum potassium >5.5 mmol/L
4. Abnormal LFTs (i.e. serum transaminases >2x ULN)
5. Sitting SBP >180 mmHg
6. Recent (<6 months) MI, CVA, TIA, revascularisation procedure
7. Ethanol abuse (in the opinion of the investigator)
8. Concomitant drug therapy that may impact on BP e.g. NSAIDs, COX-2 inhibitors, other antihypertensive agents
9. Unable to comply with study requirements (in the opinion of the investigator)
10. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure between the groups | 12 weeks

SECONDARY OUTCOMES:
Absolute cardiovascular risk | 12 weeks
  Measurements will be performed at baseline and 12 weeks of key variables that contribute to absolute cardiovascular risk.
Safety parameters | 12 weeks
  Frequency of drug-related adverse events and major cardiovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia